CLINICAL TRIAL: NCT05269368
Title: Intérêt du méchage Pour la Chirurgie Ossiculaire et la Myringoplastie : Essai contrôlé randomisé Multicentrique de Non-infériorité
Brief Title: Interest of Wicking for Ossicular Surgery and Myringoplasty
Acronym: MECH-ORL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DR210132-MECH-ORL; 2021-A02788-33 (Registry Identifier: Id-RCB-ANSM-France); 221 A15 (Other: Comité de Protection des Personnes Sud-Méditerranée II)
Record Dates: First submitted 2022-01-21; First posted 2022-03-08 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Post-Op Complication; Otologic Disease
Keywords: Ossicular surgery; Otological surgeries; Wicking
MeSH Terms: conditions — Postoperative Complications; Ear Diseases | interventions — Capillary Action

STUDY DESIGN:
Intervention Model Description: * Experimental group: No Wicking
  * Control groupe: Wicking after intervention
Who Masked: Outcomes Assessor
Masking Description: Three experts, independent of the study, will examine the photos three months after the intervention using a standardized evaluation grid based on 10 criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No wicking (Experimental): Absence of Wicking after intervention
  Interventions: Procedure: No wicking
- Control (Active Comparator): Wicking after intervention
  Interventions: Procedure: Wicking

INTERVENTIONS:
Procedure: Wicking — Absorbable or non-absorbable wicking
  Arms: Control
Procedure: No wicking — No wicking after surgery
  Arms: No wicking

SUMMARY:
Myringoplasties and ossicular surgery are very common procedures. Following these otological surgeries, most surgeons install a wicking. This intervention consists of placing a wick, absorbable or not, in the external acoustic meatus, after having replaced the tympanomeatal flap.

DETAILED DESCRIPTION:
Myringoplasties and ossicular surgery are very common procedures. Following these otological surgeries, most surgeons install a wicking. This intervention consists of placing a wick, absorbable or not, in the external acoustic meatus, after having replaced the tympanomeatal flap.

Putting in place a wicking often requires to remove this wicking, feared by the patient. In addition, wicking leads to obstruction of the external acoustic meatus responsible for functional discomfort (feeling of fullness in the ear, pain, significant conductive deafness) which can last from one to several weeks depending on the type of wicking.

Despite these drawbacks, the rationale for wicking has never been established, the choice of wick type is often empirical, and its necessity is sometimes controversial in the literature. Recent studies have studied the absence of wicking as an alternative to overcome its many drawbacks. No prospective, randomized, multicenter study has been performed to show the superiority of wicking in healing following middle ear surgery (myringoplasty, stapedo-vestibular ankylosis, ossiculoplasty) via the duct or the endaural route. The only study with a high level of evidence concerns only endoscopic surgery. This study has the advantage of showing that with comparable audiometric and healing results, the absence of wicking allows a reduced operating time, an earlier reduction in otorrhea and the feeling of blocked ears, and an earlier improvement of hearing. Given this work in the literature, our hypothesis is that tympanic healing is not impaired in the absence of wicking.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age 18 = or + ), whose mother tongue is French or who understands French language
* Ossicular surgery (fitting of a partial or total ossicular prosthesis) or myringoplasty performed endoscopically, from the speculum, from the duct or from the endaural.
* Tympanic reconstruction by all types of grafts: cartilage, fascia, autologous fat
* Written consent signed by the participant
* Affiliation to a social security scheme,

Exclusion Criteria:

* Pregnant or breastfeeding woman, patient under legal protection, guardianship or curatorship.
* Need for a retroauricular approach.
* Need for annulus detachment> 60%
* Presence of cholesteatoma or middle ear tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2025-05-16 (Estimated); Study Completion 2026-05-16 (Estimated)

PRIMARY OUTCOMES:
Tympanic and external auditory canal healing | Three months after intervention.
  Healing of tympanic membrane and external auditory canal, evaluated blindly by 3 experts, on an oto-endoscopy picture.

SECONDARY OUTCOMES:
Audiometric results | Pre-operative, 3 months, 12 months
  Audiometric results defined by the pure-tone average on 500, 1000, 2000 and 3000 Hz frequencies.
Post-operative satisfaction | Immediate post-operative, day 7-10, day 30, 3 months
  Visual Analogic scale (0-10 (min-max))
Post-operative pain | Immediate post operative,day 7-10, day 30, 3 months
  Visual Analogic scale (0-10 (min-max))
Post-operative quality of life | Day 7-10, day 30, 3 months,12 months
  Glasgow Benefit Inventory (-100 (min) to +100 (max))
Post-operative stress | Pre-operative, day 7-10, day 30, 3 months, 12 months
  Perceived Stress Scale (PSS-10) 10-50 (min-max) Never to often
Operative time | 30-120 minutes
  Operative time of the otology surgery, in minutes
Complications | At any time of the follow-up,up to 1 year
  Questionnaire given to surgeons, allowing description of complications

CONTACTS AND LOCATIONS:
Overall Officials: Charles AUSSEDAT, MD, Study Director — University Hospital of TOURS
Locations (6):
- France (6):
  - Hospital Blois, Blois
  - University Hospital BREST, Brest
  - Hospital Le Mans, Le Mans
  - University Hospital NANTES, Nantes
  - Hospital La Pitié Salpêtrière-APHP, Paris
  - University Hospital TOURS, Tours

IPD SHARING:
Plan to Share IPD: No